CLINICAL TRIAL: NCT03653520
Title: Conscious Sedation Efficacy of the Novel Medication, MKO Melt (Midazolam, Ketamine, Ondansetron), During Cataract Surgery
Brief Title: Conscious Sedation Efficacy of the MKO Melt (Midazolam, Ketamine, Ondansetron)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Avanti Anesthesia (Other)
Responsible Party: Principal Investigator, Maggie Jeffries, Principal Investigator, Avanti Anesthesia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ANES001
Record Dates: First submitted 2018-08-23; First posted 2018-08-31 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract | interventions — Diazepam; Tramadol; Ondansetron

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: The surgeon was not aware which medication the patient received
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- diazepam only (group 1) (Active Comparator): Patients are given 5 or 10mg of diazepam for sedation before surgery for sedation
  Interventions: Drug: Diazepam
- diazepam/tramadol/ondansetron (group 2) (Active Comparator): Patients are given 5 or 10mg of diazepam, 50 or 100mg of tramadol and 4 or 8mg of ondansetron orally before surgery for sedation
  Interventions: Drug: Diazepam; Drug: Tramadol; Drug: Ondansetron
- MKO only (group 3) (Experimental): Patients are given 1 or 2 MKO melts (each contain 3mg midazolam, 25mg ketamine, 2mg ondansetron) sublingually before surgery for sedation
  Interventions: Drug: MKO melt

INTERVENTIONS:
Drug: Diazepam — 5 or 10mg
  Arms: diazepam only (group 1); diazepam/tramadol/ondansetron (group 2)
Drug: Tramadol — 50mg or 100mg
  Arms: diazepam/tramadol/ondansetron (group 2)
Drug: Ondansetron — 1 or two tabs
  Arms: diazepam/tramadol/ondansetron (group 2)
Drug: MKO melt — 1 or 2 MKO melts
  Arms: MKO only (group 3)

SUMMARY:
The investigators hypothesized that the combination of Valium, Tramadol and Zofran is superior to the substantially more expensive MKO melt in patient satisfaction after cataract surgery.

DETAILED DESCRIPTION:
The MKO melt is being marketed as an anesthetic medication for cataract surgery that has the advantage that it eliminates the need for an IV in 85% of patients although that number was established anecdotally. This alternative, however, is very cost limiting.The investigators wanted to see if the current regimen (valium only) or a combination similar to the MKO melt (valium + tramadol + zofran) are as good if not better than the MKO melt for anesthesia and how many patients could have indeed gone with an intravenous line (didn't need any extra medications).

ELIGIBILITY:
Inclusion Criteria:

* All patients scheduled to undergo cataract surgery with Drs. Mayo and Wade at Kirby Glen Surgery Center

Exclusion Criteria:

* Age <18 years
* Patient is not suitable for the medications for reasons such as unsteady gait, cane, wheelchair, severe dementia (unable to consent), terminal illness
* Allergy to a medication in protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 651 (Actual)
Dates: Start 2017-06-28 (Actual); Primary Completion 2017-11-02 (Actual); Study Completion 2017-11-04 (Actual)

PRIMARY OUTCOMES:
Number of patient who needed additional IV medication for cataract surgery | 1 day
  Patients who require IV medications for self-reported pain or anxiety during surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Maggie Jeffries, MD, Principal Investigator — Avanti Anesthesia
Locations (1):
- Memorial Hermann Kirby Glen Surgery Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
De-identified individual participant data for all primary and secondary outcome measures will be available to those who contact primary investigator. We may decide to fully publish data but are undecided.

DOCUMENTS (2):
  • Study Protocol (2017-04-03): https://cdn.clinicaltrials.gov/large-docs/20/NCT03653520/Prot_000.pdf
  • Informed Consent Form (2017-04-03): https://cdn.clinicaltrials.gov/large-docs/20/NCT03653520/ICF_001.pdf